CLINICAL TRIAL: NCT01495026
Title: An Open-label, Randomized, Single Dose, Multi-stage, Cross-over Study to Determine the Relative Bioavailability of Fixed Dose Combination Products Containing a 3-oblong Dutasteride Soft Gel Capsule and Tamsulosin (0.5 mg Dutasteride /0.2 mg Tamsulosin HCl) Pellets Having a Range of Tamsulosin Release Rates Produced by Different Mixtures of Enteric Coated and Uncoated Pellets Relative to Harnal-D Tablets, in Healthy Male Subjects of North East Asian Ancestry.
Brief Title: A Study Assessing a Range of Formulations of the Fixed Dose Combination Product Containing Dutasteride (0.5mg) and Tamsulosin Hydrochloride (0.2mg) to Find a Formulation Which is Bioequivalent to Harnal-D Tablets (Tamsulosin Hydrochloride, 0.2mg) in Healthy Male Subjects From North East Asia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 115708
Record Dates: First submitted 2011-12-15; First posted 2011-12-19 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Prostatic Hyperplasia
Keywords: Healthy male subjects; North-East Asian ancestry; Bioequivalence; Food effect; Tamsulosin hydrochloride; Cross-over design; Pilot bioequivalence; Dutasteride (GI198745)
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Dutasteride; Tamsulosin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Fixed dose combination product (Experimental): Fixed dose combination capsule containing dutasteride 0.5mg and tamsulosin 0.2mg
  Interventions: Drug: Dutasteride (0.5mg, fasted state); Drug: Dutasteride (0.5mg, fed state); Drug: Harnal-D Tablets with water (fasted state); Drug: Harnal-D Tablets with water (fed state); Drug: Harnal-D tablets without water (fasted state)
- Dutasteride (Experimental): Commercial formulation of Dutasteride 0.5mg
  Interventions: Drug: Fixed dose combination capsule containing dutasteride 0.5mg and tamsulosin 0.2mg (fasted state); Drug: Fixed dose combination capsule containing dutasteride 0.5mg and tamsulosin 0.2mg (fed state)
- Harnal-D Tablets (Experimental): Commercial formulation of Harna--D Tablets comprising 0.2mg Tamsulosin Hydrochloride
  Interventions: Drug: Dutasteride (0.5mg, fasted state); Drug: Dutasteride (0.5mg, fed state); Drug: Fixed dose combination capsule containing dutasteride 0.5mg and tamsulosin 0.2mg (fasted state); Drug: Fixed dose combination capsule containing dutasteride 0.5mg and tamsulosin 0.2mg (fed state)

INTERVENTIONS:
Drug: Dutasteride (0.5mg, fasted state) — Open-label, randomized, single dose, multi-stage, cross-over study
  Arms: Fixed dose combination product; Harnal-D Tablets
Drug: Dutasteride (0.5mg, fed state) — Commercial formulation of Dutasteride 0.5mg
  Arms: Fixed dose combination product; Harnal-D Tablets
Drug: Fixed dose combination capsule containing dutasteride 0.5mg and tamsulosin 0.2mg (fasted state) — FDC with 85%, 65% and 0% of the dose as enteric-coated pellets and with X and/or Y% of the dose as enteric-coated pellets (X and Y to be determined from PK results from Stage 1)
  Arms: Dutasteride; Harnal-D Tablets
Drug: Fixed dose combination capsule containing dutasteride 0.5mg and tamsulosin 0.2mg (fasted state) — FDC containing faster-release enteric-coated pellets
  Arms: Dutasteride; Harnal-D Tablets
Drug: Fixed dose combination capsule containing dutasteride 0.5mg and tamsulosin 0.2mg (fasted state) — FDC bioequivalent to Harnal-D tablets
  Arms: Dutasteride; Harnal-D Tablets
Drug: Fixed dose combination capsule containing dutasteride 0.5mg and tamsulosin 0.2mg (fed state) — FDC bioequivalent to Harnal-D tablets
  Arms: Dutasteride; Harnal-D Tablets
Drug: Harnal-D Tablets with water (fasted state) — Commercial formulation of Harnal-D Tablets
  Arms: Fixed dose combination product
Drug: Harnal-D Tablets with water (fed state) — Commercial formulation of Harnal-D Tablets
  Arms: Fixed dose combination product
Drug: Harnal-D tablets without water (fasted state) — Commercial formulation of Harnal-D Tablets
  Arms: Fixed dose combination product

SUMMARY:
This study is an open-label, randomized, single dose, multi-stage, cross-over study in healthy male subjects of North East Asian ancestry. The aims are to:

* evaluate the pharmacokinetic parameters of several formulations of a fixed dose combination (FDC) capsule of dutasteride and tamsulosin hydrochloride (0.5 mg/0.2 mg) relative to co-administration of dutasteride 0.5 mg capsules and tamsulosin hydrochloride 0.2 mg tablets in the fasted state in order to define a formulation which is bioequivalent to a 0.2 mg orally disintegrating tamsulosin tablet, (Harnal-D Tablets)
* determine the effect of food on the relative bioavailability of tamsulosin in the FDC product which is assessed to be bioequivalent to Harnal-D Tablets in the fasted state
* assess the effect of water on the relative bioavailability of tamsulosin in Harnal-D Tablets in the fasted state
* assess the safety and tolerability of dosing with the different FDC capsule formulations Subjects will receive single oral doses in at least one treatment period; treatment periods will be separated by a 5-10 day washout period. Blood samples for pharmacokinetic analysis will be taken at regular intervals after dosing. Safety will be assessed by measurement of blood pressure, heart rate and review of adverse events. Each stage of the study will enrol 18 subjects to ensure 16 complete. Subjects may consent to participate in more than one stage.

DETAILED DESCRIPTION:
This study is an open-label, randomized, single dose, multi-stage, cross-over study in healthy male subjects of North East Asian ancestry. The aims are to:

* evaluate the pharmacokinetic parameters of several formulations of a fixed dose combination (FDC) capsule of dutasteride and tamsulosin hydrochloride (0.5 mg/0.2 mg) relative to co-administration of dutasteride 0.5 mg capsules and tamsulosin hydrochloride 0.2 mg tablets in the fasted state in order to define a formulation which is bioequivalent to a 0.2 mg orally disintegrating tamsulosin tablet, (Harnal-D Tablets)
* determine the effect of food on the relative bioavailability of tamsulosin in the FDC product which is assessed to be bioequivalent to Harnal-D Tablets in the fasted state
* assess the effect of water on the relative bioavailability of tamsulosin in Harnal-D Tablets in the fasted state
* assess the safety and tolerability of dosing with the different FDC capsule formulations Subjects will receive single oral doses in at least one treatment period; treatment periods will be separated by a 5-10 day washout period. Blood samples for pharmacokinetic analysis will be taken at regular intervals after dosing. Safety will be assessed by measurement of blood pressure, heart rate and review of adverse events. Each stage of the study will enrol 18 subjects to ensure 16 complete. Subjects may consent to participate in more than one stage.

BACKGROUND:

Dutasteride:

Dutasteride (AVODART ™) is an approved potent 5-alpha-reductase inhibitor indicated for the treatment of symptomatic benign prostatic hyperplasia (BPH) in men with an enlarged prostate to improve symptoms, reduce the risk of acute urinary retention and reduce the risk of the need for BPH-related surgery [AVODART Package Insert, 2009]. In humans, dutasteride is well-tolerated in single doses up to 40mg/day, multiple doses up to 40mg/day administered for 7 days, and 5 mg/day administered for 24 weeks. In single dose clinical studies, the overall incidence and type of adverse events (AEs) was similar across the dutasteride, placebo, and finasteride treatment groups.

Tamsulosin:

Tamsulosin (Harnal, Harnal D, Flomax) is an alpha-1-adrenoceptor blocking agent approved for the treatment of signs and symptoms of benign prostatic hyperplasia. Tamsulosin HCl is extensively metabolized, with less than 10% of the dose excreted in the urine unchanged [Harnal, 2009; Harnal, 2011; Flomax, 2011]. In human liver microsomes and human lymphoblastoid cells expressing CYP cDNAs in vitro, tamsulosin HCl is metabolized by both CYP3A4 and CYP2D6 [Matsushima, 1998].

Dutasteride and Tamsulosin:

Clinical data exist to support that tamsulosin (an alpha-1-adrenoceptor antagonist), when used in combination with dutasteride (a 5-alpha reductase inhibitor), offers a more effective treatment for the symptoms of benign prostatic hyperplasia than either drug used alone [GSK study ARI40005, GlaxoSmithKline document number HM2002/00171/01]. In addition, data from a large, multi-centre National Institutes of Health-sponsored Medical Therapy of Prostatic Symptoms (MTOPS) study revealed greater benefits of combination alpha-1-adreoceptor antagonist and 5-alpha-reductase inhibitor therapy compared with either monotherapy in males with BPH [McConnell, 2002]. Clinical drug interaction studies have shown no pharmacokinetic or pharmacodynamic interactions between dutasteride and tamsulosin. Dutasteride may be administered with or without food. Tamsulosin should be administered with food.

Food effect PK data exists for co-administration of dutasteride and tamsulosin given in a fixed dose combination (FDC) capsule formulation relative to the co-administration of the two components, dutasteride and tamsulosin HCl; GSK studies ARI109882, [GlaxoSmithKline document number ZM2007/00022/00], and ARI114694, [GlaxoSmithKline document number ZM2010/00028/00]. In the latter study, the dose of tamsulosin HCl administered was 0.2 mg versus 0.4mg administered in ARI109882. The dose of dutasteride was the same in both studies (0.5mg). In ARI109882, the GSK combination capsule was found to be bioequivalent (under both fed and fasted conditions) to the marketed products administered separately. ARI114694 demonstrated bioequivalence for dutasteride but not for tamsulosin when administered as an FDC product (of dutasteride 0.5 mg and tamsulosin 0.2 mg) relative to co-administration of separate commercial formulations of dutasteride (0.5 mg) and tamsulosin (0.2 mg) in the fed and fasted stage in different North East Asian ethnic groups.

A subsequent GSK study, ARI115707, therefore investigated the relative bioavailability of tamsulosin (0.2mg tamsulosin HCl) only in the FDC product. Two different enteric-coated formulations of tamsulosin were administered with a 3-oblong dutasteride soft gel (0.5 mg) as a FDC capsule relative to co-administration of Harnal Capsules or Harnal-D Tablets with unbranded AVODART (0.5mg dutasteride). The two FDC formulations consisted of: 10% (weight gain) enteric coated tamsulosin pellets with a 3-oblong dutasteride soft gel and 15% (weight gain) enteric coated tamsulosin pellets with a 3-oblong dutasteride soft gel. Specifically, the study aimed to investigate the relative bioavailability of the following:

* FDC (with 10% enteric coated tamsulosin pellets) to a commercial formulation of dutasteride plus tamsulosin (Harnal-D Tablet)
* FDC (with 10% enteric coated tamsulosin pellets) to a commercial formulation of dutasteride plus tamsulosin (Harnal Capsule)
* FDC (with 15% enteric coated tamsulosin pellets) to a commercial formulation of dutasteride plus tamsulosin (Harnal-D Tablet) (also investigated in ARI114694)
* FDC (with 15% enteric coated tamsulosin pellets) to a commercial formulation of dutasteride plus tamsulosin (Harnal Capsule).

ARI115707 results showed that the GSK combination capsule with 10% enteric coated tamsulosin pellets was bioequivalent to the Harnal Capsule. None of the two GSK formulations was found to be bioequivalent to the Harnal-D Tablet.

In this study ARI115708, the relative bioavailability of tamsulosin (0.2mg tamsulosin HCl) is further investigated in several different formulations administered with a 3-oblong dutasteride soft gel as a FDC capsule relative to co-administration of Harnal-D Tablets (0.2 mg) with unbranded AVODART (dutasteride, 0.5mg). All formulations will be administered in the fasted state except in the last stage where the effect of food on the FDC will be assessed as well as the effect of water on the administration of Harnal-D Tablets. As Harnal Capsules are not available in Korea or Japan, bioequivalence to Harnal-D Tablets would allow the FDC to be registered in China, Korea, Taiwan and Japan, where Harnal-D Tablets are approved. Therefore, in ARI115708, only Harnal-D Tablets are used as the comparator.

ELIGIBILITY:
Inclusion Criteria:

A subject will be eligible for inclusion in this study only if all of the following criteria apply:

* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Males between 20 and 45 years of age inclusive, at the time of signing the informed consent form.
* Japanese ancestry defined as being born in Japan, having four ethnic Japanese grandparents, holding a Japanese passport or identity papers and being able to speak Japanese, or Korean ancestry defined as being born in Korea, having four ethnic Korean grandparents, holding a Korean passport or identity papers and being able to speak Korean, or Chinese ancestry defined as being born in China, Hong Kong, Singapore or Taiwan, having four ethnic Chinese grandparents, holding a Chinese passport or identity papers and being able to speak Chinese.

Japanese, Korean and Chinese subjects should also have lived outside their respective countries for less than 10 years.

* Male subjects with female partners of child-bearing potential must agree to use one of the protocol-approved contraception methods. This criterion must be followed from the time of the first dose of study medication until 45 days after the last dose.
* BMI within the range 18 -28 kg/m2 (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Single QTc < 450 msec; or QTc < 480 msec in subjects with Bundle Branch Block.
* AST, ALT, alkaline phosphatase and bilirubin less than or equal to 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).

Exclusion Criteria:

A subject will not be eligible for inclusion in this study if any of the following criteria apply:

Medical Condition Exclusions:

* Poor metabolizer for CYP2D6 substrates as determined by genotyping of selected CYP2D6 variants at screening.
* History of postural hypotension, dizziness, poor hydration, vertigo, vaso-vagal reactions or any other signs and symptoms of orthostasis, which in the opinion of the investigator could be exacerbated by tamsulosin and result in putting the subject at risk of injury.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* A positive test for HIV antibody.

Medical Exclusions:

* Subjects must be able and willing to refrain from use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort, Black Khosh, Dong Quai, Milk Thistle, licorice) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of sensitivity to tamsulosin HCl or dutasteride, components thereof or drugs of this class or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* A history of sensitivity to heparin or heparin-induced thrombocytopenia
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.

Lifestyle Exclusions:

* A positive pre-study drug/alcohol screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines.
* History of regular alcohol consumption within 6 months of the screening visit defined by the following Australian guidelines:

Males: An average weekly intake greater than 21 units or an average daily intake greater than 3 units. One unit is equivalent to 270 mL of full strength beer, 470 mL of light beer, 30 mL of spirits and 100 mL of wine.

Subjects must be able and willing to abstain from beverages and foods containing alcohol 24 hours prior to and during the dosing day.

* Consumption of red wine, grapefruit juice, grapefruit and related hybrids from 7 days prior to the first dose of study medication.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2011-11-06 (Actual); Primary Completion 2012-04-03 (Actual); Study Completion 2012-04-03 (Actual)

PRIMARY OUTCOMES:
Relative bioavailability of tamsulosin from FDC products (0.5 mg dutasteride /0.2 mg tamsulosin HCl) containing a size 3-oblong dutasteride soft gel capsule and tamsulosin pellets having a range of tamsulosin release rates produced by different mixtures | 0, 15 min, 30 min, 45 min, 1 hr, 2 hr, 3 hr, 4 hr, 6 hr, 8 hr, 10 hr, 12 hr, 16 hr, 24 hr, 48 hr, 72 hr

SECONDARY OUTCOMES:
Effect of food on the relative bioavailability of tamsulosin in a selected FDC product in healthy male subjects of North East Asian ancestry | 0, 15 min, 30 min, 45 min, 1 hr, 2 hr, 3 hr, 4 hr, 6 hr, 8 hr, 10 hr, 12 hr, 16 hr, 24 hr, 48 hr, 72 hr
Effect of water on the relative bioavailability of tamsulosin in Harnal-D Tablets in the fasted state in healthy male subjects of North East Asian ancestry. | 0, 15 min, 30 min, 45 min, 1 hr, 2 hr, 3 hr, 4 hr, 6 hr, 8 hr, 10 hr, 12 hr, 16 hr, 24 hr, 48 hr, 72 hr
Safety and tolerability of dosing with the different FDC capsule formulations in healthy male subjects of North East Asian ancestry | Vital signs: 0, 2 hr, 4 hr, 6 hr, 10 hr, 24 hr, 48 hr and 72 hr. Adverse events: 5 timepoints from pre-dose to follow-up visit (10-14 days post-dose)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Randwick, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] AVODART (Dutasteride 0.5 mg) Product Information. March 2011.
- [Background] Cai G, Thiessen JJ, Baidoo CA, Fossler MJ. Operating characteristics of a partial-block randomized crossover bioequivalence study for dutasteride, a drug with a long half-life: investigation through simulation and comparison with final results. J Clin Pharmacol. 2010 Oct;50(10):1142-50. doi: 10.1177/0091270009355155. Epub 2010 Feb 16. PMID 20160156
- [Background] FLOMAX (Tamsulosin hydrochloride) Product Information. January, 2011.
- [Background] Food and Drug Administration (FDA). Guidance for Industry: Handling and Retention of BA and BE Testing Samples. Centre for Drug Evaluation and Research, USA; 2004.
- [Background] GlaxoSmithKline Document Number HM2002/00171/01 Study ID ARI40005. A randomised, double-blind, parallel group study to investigate the efficacy and safety of treatment with Dutasteride (0.5mg) and Tamsulosin (0.4mg), administered once daily for 4 years, alone and in combination, on the improvement of symptoms and clinical outcome in men with moderate to severe symptomatic benign prostatic hyperplasia;. Report Date 09-Jul-2004.
- [Background] GlaxoSmithKline Document Number ZM2008/00126/02. Dutasteride Clinical Investigators Brochure v10. Report Date 27 May 2011.
- [Background] HARNAL (Tamsulosin hydrochloride 0.2 mg) Product Information. , 2011.
- [Background] HARNAL-D (Tamsulosin hydrochloride 0.2 mg) Product Information. , 2009.
- [Background] Matsushima H, Kamimura H, Soeishi Y, Watanabe T, Higuchi S, Tsunoo M. Pharmacokinetics and plasma protein binding of tamsulosin hydrochloride in rats, dogs, and humans. Drug Metab Dispos. 1998 Mar;26(3):240-5. PMID 9492387
- [Background] McConnell JD. The long term effects of medical therapy on the progression of BPH: Results from the MTOPS Trial (abstract 1042). 167 (4):265, 2002. J. Urology. 2002;167 (4):265.
- [Background] Schuirmann DJ. A comparison of the two one-sided tests procedure and the power approach for assessing the equivalence of average bioavailability. J Pharmacokinet Biopharm. 1987 Dec;15(6):657-80. doi: 10.1007/BF01068419. PMID 3450848
- [Result] GlaxoSmithKline Document Number 2011N112801_00 Study ID ARI114694. GlaxoSmithKline studyARI114694: An open-label, randomized, single dose, two-period cross-over study to determine the bioavailability of a fixed dose combination capsule formulation of dutasteride and tamsulosin hydrochloride (0.5 mg/0.2mg) relative to co-administration of dutasteride 0.5mg capsules and tamsulosin hydrochloride 0.2mg tablets in healthy male subjects of north east Asian and non-Asian ancestry;. Report Date 02-May-2011.
- [Result] GlaxoSmithKline Document Number RM2001/00128/01 Study ID ARI10019. A Double-Blind, Placebo Controlled, Randomized, Parallel Group Study To Investigate The Changes In The Corrected QT Interval Following Repeat Oral Doses Of GI198745 In Healthy Male Volunteers. Report Date 02-Oct-2002.
- [Result] GlaxoSmithKline Document Number RM2003/00174/01 Study ID ARI10021. An Open-Label, Single Dose, 2-Way Cross-over Study to Investigate the Pharmacokinetics, Safety and Tolerability of oral Flomax (tamsulosin hydrochloride 0.4mg capsule-US) and Omnic (tamsulosin hydrochloride 0.4mg capsule-Germany) in Healthy Male Volunteers. Report Date 04-Sep-2003.
- [Result] GlaxoSmithKline Document Number ZM2007/00022/00 Study ID ARI109882. An Open-Label, Randomized, Single Dose, Three-Period Cross-over Study to Determine the Bioequivalence and Food Effect of a Combination Capsule Formulation of Dutasteride and Tamsulosin Hydrochloride (0.5mg/0.4mg) Compared to Concomitant Dosing of AVODART 0.5mg and FLOMAX 0.4 mg Commercial Capsules in Healthy Male Subjects. Report Date 30-Aug-2007.
- See also: Results for study 115708 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/115708?search=study&search_terms=115708#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 115708 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 115708 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 115708 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 115708 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 115708 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 115708 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 115708 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register